CLINICAL TRIAL: NCT01429623
Title: A 36-month, Multi-centre, Randomized, Double Blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of Low Dose Ladostigil in Patients With Mild Cognitive Impairment (MCI)
Brief Title: A 3 Year Study to Evaluate the Safety and Efficacy of Low Dose Ladostigil in Patients With Mild Cognitive Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avraham Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CO17730; 2011-004187-30 (EudraCT Number)
Record Dates: First submitted 2011-09-03; First posted 2011-09-07 (Estimated); Results first posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Mild Cognitive Impairment; Dementia
Keywords: Mild Cognitive Impairment; Early Stage Dementia; Conversion to Alzheimer's disease; Memory Impairment
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Memory Disorders | interventions — (N-propargyl-(3R) aminoindan-5-yl)-ethyl methyl carbamate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ladostigil hemitartrate (Experimental): 10mg ladostigil base
  Interventions: Drug: ladostigil hemitartrate
- Placebo Control (Placebo Comparator): drug product excipients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ladostigil hemitartrate — 10mg ladostigil base administered once daily as hard gelatin capsule
  Other Names: ladostigil; Ladostigil capsules
  Arms: ladostigil hemitartrate
Drug: Placebo — Placebo comparator
  Arms: Placebo Control

SUMMARY:
The purpose of this study is to determine whether treatment with the investigational drug ladostigil will delay the onset of Alzheimer's disease(AD) in patients with Mild Cognitive Impairment (MCI). MCI is now recognized as a precursor to AD and clinical tools are available to assess cognitive performance at this earlier stage. Ladostigil is currently under investigation for the treatment of AD. In this study, the investigators will be examining ladostigil at a lower dose level. At this dose level, ladostigil has been shown to reduce signs of early memory loss in animals. Thus, in this study the investigators are attempting to determine if earlier invention with a lower dose of ladostigil will significantly reduce initial memory loss and delay the subsequent progression to more serious cognitive dysfunction.

DETAILED DESCRIPTION:
Ladostigil shows neuroprotective activity, reducing oxidative stress, activating microglia, and inhibiting pro-inflammatory cytokines in pre-clinical models. Study assessed its safety and potential efficacy in a 3-year, randomised, double-blind, placebo-controlled, phase 2 clinical trial in patients with mild cognitive impairment (MCI). Patients from 16 centers in Austria, Germany and Israel with MCI (Albert et al 2011), Clinical Dementia Rating (CDR) = 0.5, Mini-Mental State Examination (MMSE) > 24, Wechsler Memory Scale - Revised Verbal Paired Associates ≤ 18, and medial temporal lobe atrophy were stratified by APOE4 genotype and randomly assigned (1:1 allocation) using blocks of 4, to receive either ladostigil, 10 mg per day, or placebo as identically-appearing capsules. The primary endpoint was onset of Alzheimer's disease (AD). Secondary endpoints were the NTB, DAD, and GDS. Exploratory outcomes were MRI-derived whole brain, hippocampus, and entorhinal cortex volumes; the NeuroTrax Mindstreams computerized cognitive battery; and the CDR. Between February 17, 2012 and August 1, 2013, we randomly allocated 210 patients to placebo (107 patients) or ladostigil (103 patients); 4 patients in each group lacked post baseline assessments. After 36 months 20.4% (21 of 103 patients) of the placebo group and 14.1% (14 of 99 patients) of the ladostigil group progressed to AD (log-rank test p=.16). There were no significant effects on NTB, DAD, or GDS outcomes. There was less decline in whole brain volume in the ladostigil group as compared to placebo (p<.02), but not hippocampus and entorhinal cortex volumes, and CDR and a trend for less decline on the RAVLT total delayed score component of the NTB (p=.09). Fourteen patients taking placebo and 21 taking ladostigil discontinued treatment because of adverse events. Serious adverse events were reported by 26 (25.2%) patients in the ladostigil group and 28 (26.2%) patients in the placebo group. Ladostigil appeared safe, well-tolerated, and may have potential for improving memory and delaying progression to dementia.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (non-childbearing potential) with a diagnosis of Mild Cognitive Impairment (MCI) according to consensus criteria as defined by Petersen
* Abnormal memory function will be evaluated by Verbal Paired Associates from the Wechsler Memory Scale - Revised. Norm values for healthy adults in two age cohorts are: a) 50-70 years 19.7 (SD=2.9) and b) 75-95 years 18.3 (SD=2.8). Patients that score < or = 23 will be included.
* Clinical Dementia Rating (CDR) score of 0.5 (Memory box score 0.5 or 1, no box score > 1)
* Mini Mental State Examination (MMSE) > 24 and < or = 30
* General cognition and functional performance is sufficiently preserved such that a diagnosis of AD can be excluded by the site physician at the time of the screening visit.
* No significant cerebrovascular disease indicated by Modified Hackinski Ischaemic Score equal to or below 4
* Age 55-85 years based upon correlation of cognition and Scheltens score observed in this age range
* Geriatric Depression Scale (GDS) of < or = 5
* An informer who has frequent contact with the subject (e.g. an average of 10 hours per week or more) is available and agrees to monitor administration of study drug, to observe the subject for adverse events and to accompany the subject to clinical visits during the trial, if the presence of the informer is required.
* All patients have to undergo an MRI scan after the screening visit, i.e. during the screening visit, irrespective of MRIs having been performed prior to entry into the study. MRI findings have to be consistent with a diagnosis of MCI.
* Central rating of medial temporal lobe according to Scheltens scale. The right and left medial temporal structures will be rated separately and an overall estimate will be deduced using the average of the two ratings. An average score > 1 is required to make patients eligible for the study.
* Adequate visual and auditory acuity must be demonstrated to allow for neuropsychological testing.
* Good general health status acceptable for participation in a 36-month clinical trial, with no additional diseases expected to interfere with the study
* ECG without clinically significant abnormalities according to exclusion criteria listed below
* Subject is not pregnant, lactating or of childbearing potential (i.e. women must be two years post menopausal or surgically sterile)
* Signed informed consent by patient and informer prior to any study specific procedure

Exclusion Criteria:

* Failure to perform screening or baseline examinations
* Any significant neurological disease other than suspected MCI
* MRI exclusion criteria which allow for mild concomitant vascular lesions are:

  * Thromboembolic infarction
  * Other focal lesions which may be responsible for the cognitive status of the patient such as infectious disease, space-occupying lesions, normal pressure hydrocephalus or any other abnormalities associated with significant central nervous disease
  * More than one lacunar infarct defined as a focal lesion of CSF signal intensity with a diameter of < 1.5cm in any dimension
  * Any lacunar infarct in a strategically important location such as the thalamus, hippocampus of either hemisphere, head of the left caudate
  * White matter lesions involving more than 25% of the hemispheric white matter
  * Implants such as pacemakers, insulin pumps, cochlear implants, nerve stimulators, implantable cardioverter defibrillators, and other medical implants that have not been certified for MRI
  * Ferromagnetic foreign bodies such as shell fragments need to be considered on an individual basis
  * Metallic implants that can cause artifacts and RF induced heating such as surgical prostheses or aneurysm clips need to be considered on an individual basis
* Clinical or laboratory findings consistent with:

  * Central nervous system diseases such as those resulting from severe head trauma, tumours, subdural haematomas or other space occupying processes, etc
  * Seizure disorder
  * Other infectious, metabolic or systemic diseases affecting central nervous system (syphilis, present hypothyroidism, present vitamin B12 or folate deficiency, serum electrolytes out of normal range, juvenile onset diabetes mellitus, etc)
* History or evidence of schizophrenia or bipolar disorder (DSM IV criteria); active major depression
* Clinically significant advanced or unstable disease that may interfere with primary or secondary variable evaluations, and which may bias the assessment of the clinical or mental status of the patient or put the patient at special risk, such as:

  * Malignant tumours within the last five years except skin malignancies (other than melanoma) or indolent prostate cancer
  * Metastases
  * History of myocardial infarction within one year prior to screening or unstable or severe cardiovascular disease including angina or congestive heart failure with symptoms at rest
  * Uncontrolled hypertension (systolic pressure > 170mmHg or diastolic pressure > 100mmHg)
  * Bradycardia (persistent heart beat < 50/min) or tachycardia ( persistent heart beat > 100/min)
  * AV block (type II / Mobitz II and type III), congenital long QT syndrome, sinus node dysfunction or prolonged QTcB-interval (males > 450msec, females > 470msec)
  * Clinically significant obstructive pulmonary disease or asthma
  * Clinically significant laboratory findings that indicate abnormalities in blood biochemistry, blood haematology or urinalysis
  * Uncontrolled diabetes mellitus defined by HbA1c > 8.5
  * Clinically significant liver disease, coagulopathy or vitamin K deficiency within the past two years prior to screening
  * Renal insufficiency (serum creatinine > mg/dl or creatinine clearance < or = to 45ml/min according to Cockgroft-Gault formula); in case of creatinine clearance < or = 45ml/min, an alternative verification of the renal function must be completed using cystatin C analysis. In case of normal level of cystatin C, the patient can be included in the study.
* Any prior use of medications approved by local authorities for the treatment of Alzheimer's disease (e.g. tacrine, donepezil, rivastigmine, galantamine, memantine or other newly approved medications)
* Disability that may prevent the subject from completing all study requirements (e.g. blindness, deafness, severe language difficulty, etc)
* Women who are fertile and of child bearing potential
* Chronic daily intake of antidepressants as noted in section 9.5 of the clinical study protocol
* Suspected or known drug or alcohol abuse, i.e. more than approximately 60g alcohol (approximately 1 lter of beer or 0.5 liter of wine) per day as indicated by elevated MCV significantly above normal value at screening
* Suspected or known allergy to any components of the study treatments
* Enrollment in another investigational study or intake of investigational drug within the previous three months
* Any condition (e.g. epilepsy) which in the opinion of the investigator makes the patient unsuitable for inclusion

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2012-02; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tzvi Dwolatzky, MD, Principal Investigator — Director, Department of Geriatrics and Memory Clinic, Mental Health Center, Israel P.O. Box 4600, Beersheva 84170
Locations (12):
- Austria (3):
  - Medizinische Universitat Graz, Abteilung fur Neurologie, Graz
  - Landeskrankenhaus Hall, Memory Klinik, Hall in Tirol
  - Privatordination Rainer, Vienna
- Germany (3):
  - Studienambulanz St. Joseph Krankenhaus Berlin, Emovis GmbH, Berlin
  - Otto-von-Guericke-Universitat, Universitatsklinik fur Neurologie und fur Stereotaktische, Magdeburg
  - Studienzentrum Nordwest, Westerstede
- Israel (6):
  - Department of Geriatrics and Memory Clinic, Mental Health Center, Israel, Beersheva
  - Cognitive Neurology Unit, Rambam Health Care Campus, Haifa
  - Cognitive Clinic, Department of Geriatrics, Carmel Medical Center, Haifa
  - Department of Physical Medicine and Rehabilitation, Hadassah University Hospital, PO Box 24035, Jerusalem
  - Memory Clinic, Sheba Medical Center at Tel Hashomer, Ramat Gan
  - Center for Memory and Attention Disorders, Department of Neurology, Sourasky Medical Center, Tel Aviv

REFERENCES:
- [Background] Winblad B, Palmer K, Kivipelto M, Jelic V, Fratiglioni L, Wahlund LO, Nordberg A, Backman L, Albert M, Almkvist O, Arai H, Basun H, Blennow K, de Leon M, DeCarli C, Erkinjuntti T, Giacobini E, Graff C, Hardy J, Jack C, Jorm A, Ritchie K, van Duijn C, Visser P, Petersen RC. Mild cognitive impairment--beyond controversies, towards a consensus: report of the International Working Group on Mild Cognitive Impairment. J Intern Med. 2004 Sep;256(3):240-6. doi: 10.1111/j.1365-2796.2004.01380.x. PMID 15324367
- [Background] DeCarli C, Frisoni GB, Clark CM, Harvey D, Grundman M, Petersen RC, Thal LJ, Jin S, Jack CR Jr, Scheltens P; Alzheimer's Disease Cooperative Study Group. Qualitative estimates of medial temporal atrophy as a predictor of progression from mild cognitive impairment to dementia. Arch Neurol. 2007 Jan;64(1):108-15. doi: 10.1001/archneur.64.1.108. PMID 17210817
- [Derived] Schneider LS, Geffen Y, Rabinowitz J, Thomas RG, Schmidt R, Ropele S, Weinstock M; Ladostigil Study Group. Low-dose ladostigil for mild cognitive impairment: A phase 2 placebo-controlled clinical trial. Neurology. 2019 Oct 8;93(15):e1474-e1484. doi: 10.1212/WNL.0000000000008239. Epub 2019 Sep 6. PMID 31492718

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment between Feb. 17, 2012 and August 1, 2013.
Period: Overall Study
Arm/Group | Ladostigil Hemitartrate | Placebo Control
Started | 102 (103 allocated, 1 withdrew consent prior to first dose, 4 lacked post baseline data) | 107 (107 allocated, 4 lacked post baseline data)
Converted to Alzheimer's (Upon conversion to Alzheimer's disease, the primary endpoint, subjects removed from study) | 14 (14 of 99) | 21 (21 of 103)
Completed | 51 | 48
Not Completed | 51 | 59
Not completed — Death | 1 | 0
Not completed — Adverse Event | 7 | 14
Not completed — Withdrawal by Subject | 19 | 13
Not completed — Physician Decision | 2 | 3
Not completed — Protocol Violation | 3 | 2
Not completed — Assorted | 1 | 2
Not completed — Conversion to Alzheimer's disease | 14 | 21
Not completed — No post baseline data | 4 | 4

BASELINE CHARACTERISTICS:
Population: 103 were randomized to ladostigil, however 1 subject withdrew consent before first dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ladostigil Hemitartrate | Placebo Control | Total
Number analyzed (Participants) | 103 | 107 | 210
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 88 | 91 | 179
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (6.3) | 71.4 (6.8) | 71.35 (6.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 41 | 77
  Male | 67 | 66 | 133
Region of Enrollment [Number; unit: participants]
  Austria | 23 | 24 | 47
  Israel | 47 | 50 | 97
  Germany | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Conversion From Mild Cognitive Impairment to Alzheimer's Disease Compared to Placebo
Description: Total number of conversions from Mild Cognitive Impairment to Alzheimer's disease across entire 3 year study period. Conversion is determined, or defined, by a Clinical Dementia Rating (CDR) score of greater than or equal to one.
  Composite rating ranges from 0 no symptoms of dementia to 3 Severe symptoms of dementia.
Time Frame: 3,6,12,18,24,30 and 36 months
Population: All randomized subjects with at least one post-baseline visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Ladostigil Hemitartrate | Placebo Control
Number analyzed (Participants) | 99 | 103
Participants | 14 | 21
Statistical Analysis 1: Comparison: Ladostigil Hemitartrate vs Placebo Control; Test type: Superiority; p < 0.16, Log Rank; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.74 to 3.25]

2. Secondary Outcome: Change in Geriatric Depression Scale for Ladostigil Versus Placebo Population
Description: Mean value change (from baseline) in Geriatric Depression Scale (GDS) across entire study period. The GDS ranges from 0 to 30. Scores of 0-9 are considered "normal", 10-19 "mildly depressed", and 20-30 "severely depressed".
Time Frame: 3,6,12,18,24,30 and 36 months
Population: Modified Intent to Treat
Measure: Mean (Standard Deviation); unit: Change from basline on units on a scale
Arm/Group | Ladostigil Hemitartrate | Placebo Control
Number analyzed (Participants) | 99 | 103
Change from basline on units on a scale | .084 (1.70) | .242 (1.87)
Statistical Analysis 1: Comparison: Ladostigil Hemitartrate vs Placebo Control; Test type: Superiority; p < 0.61, Mixed Models Analysis; Mean Difference (Net) = .37, Standard Error of Mean .24

3. Secondary Outcome: Change in Neuropsychiatric Test Battery for Ladostigil Versus Placebo Population
Description: Mean value change (from baseline) in Neuropsychiatric Test Battery (NTB) across entire study period. The NTB included the following well known cognitive tests: Rey Auditory Verbal Learning Test (RAVLT), Controlled Word Association Test (COWAT), Category Fluency Test (CFT), WMS-R Digit Span, and Trail Making Part A and B. The mean value was comprised of the z score of each of these tests with all z scores in the direction of higher scores better functioning. Range -3 to +3.
Time Frame: 3,6,12,18,24,30 and 36 months
Population: Modified Intent to treat (all randomized subject with at least one post baseline assessment)
Measure: Mean (Standard Deviation); unit: Change from basline on units on a scale
Arm/Group | Ladostigil Hemitartrate | Placebo Control
Number analyzed (Participants) | 99 | 103
Change from basline on units on a scale | .21 (.55) | .17 (.43)
Statistical Analysis 1: Comparison: Ladostigil Hemitartrate vs Placebo Control; Test type: Superiority; p < 0.32, Mixed Models Analysis; Mean Difference (Net) = -0.066, Standard Error of Mean 0.085

4. Secondary Outcome: Change in Disability Assessment in Dementia for Ladostigil Versus Placebo Population
Description: Mean value change (from baseline) in Disability Assessment in Dementia (DAD) across entire study period. DAD evaluates the basic and instrumental activities in daily activities of elderly people with dementia. Higher scores reflect better functioning. DAD ranges from 0 to 100.
Time Frame: 3,6,12,18,24,30 and 36 months
Measure: Mean (Standard Deviation); unit: Change from basline on units on a scale
Arm/Group | Ladostigil Hemitartrate | Placebo Control
Number analyzed (Participants) | 99 | 103
Change from basline on units on a scale | -0.77 (8.43) | -0.40 (5.11)
Statistical Analysis 1: Comparison: Ladostigil Hemitartrate vs Placebo Control; Test type: Superiority; p < 0.97, Mixed Models Analysis; Mean Difference (Net) = .79, Standard Error of Mean 1.17

ADVERSE EVENTS:
Time Frame: 36 months
Description: Treatment emergent adverse events (i.e., occurring after first drug administration)
Arm/Group | Ladostigil Hemitartrate | Placebo Control
All-Cause Mortality (participants affected / at risk) | 1/103 | 0/107
Serious Adverse Events (participants affected / at risk) | 26/103 | 28/107
Other Adverse Events (participants affected / at risk) | 56/103 | 59/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ladostigil Hemitartrate (N=103) | Placebo Control (N=107)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) — Events rated as serious
Chest pain (General disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 4 (5)
Chronic lymphocytic leukaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Cardiac disorders) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric cancer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Metastases to peritoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Extradural abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intraocular pressure increased (Eye disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fractured coccyx (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Humerus fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lower limb fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pelvic floor muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Post polio syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rib fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung cancer metastatic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia bacterial (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gangrene (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tinea pedis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Glaucoma surgery (Surgical and medical procedures) | 2 (5) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Intraocular lens implant (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal laminectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Transurethral prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ladostigil Hemitartrate (N=103) | Placebo Control (N=107)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (10) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 6 (6) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 10 (10)
Fatigue (General disorders) | 4 (4) | 7 (8)
Nasopharyngitis (Infections and infestations) | 11 (14) | 13 (15)
Headache (Nervous system disorders) | 7 (8) | 5 (5)
Depression (Psychiatric disorders) | 6 (6) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 7 (7)
Catarct operation (Surgical and medical procedures) | 3 (4) | 7 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No